CLINICAL TRIAL: NCT00273884
Title: Phase 2 Open-Label Study of Amonafide L-Malate in Combination With Cytarabine in Subjects With Secondary Acute Myeloid Leukemia (AML)
Brief Title: Amonafide in Combination With Cytarabine in Secondary AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xanthus Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0001A3-200-GL
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2007-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Secondary AML; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — xanafide; Cytarabine

INTERVENTIONS:
Drug: Amonafide L-Malate
Drug: Cytarabine

SUMMARY:
This protocol is designed to assess the safety and efficacy of amonafide in combination with cytarabine in subjects with previously untreated secondary AML.

DETAILED DESCRIPTION:
This is a two-stage, open-label, phase 2, multicenter study of amonafide L-malate in combination with standard-dose cytarabine in subjects with secondary AML.

Amonafide is a DNA intercalating agent and inhibitor of topoisomerase II that has been extensively studied in patients with malignant solid tumors. Amonafide has also been studied in patients with AML. In three phase I clinical trials, amonafide demonstrated anti-leukemic activity, both as monotherapy and in combination with cytarabine. This protocol is designed to further assess the safety and efficacy of amonafide in combination with cytarabine in subjects with previously untreated secondary AML.

The duration of the study is approximately 42 months: enrollment approximately 18 months and subject duration up to 24 months

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of AML (≥20% blasts of myeloid lineage in bone marrow), with FAB classification other than M3, secondary to either:

  1. Known and documented exposure to prior leukemogenic chemotherapy or radiotherapy, OR
  2. Diagnosis of MDS for ≥3 months prior to study entry (prior BM slides documenting MDS must be available for central pathology review).
* Age 18 years or older.
* ECOG performance status ≤2.
* No prior induction chemotherapy for AML; at least 4 weeks since completion of prior chemotherapy for MDS. (Subjects with rapidly rising blast count may be enrolled within 4 weeks of prior cytotoxic chemotherapy).
* Fertile and sexually active men and women must use effective contraception throughout study. Women of childbearing potential must have a negative pregnancy test.
* LVEF ≥50% by MUGA or ECHO.
* Adequate renal function: serum creatinine ≤1.5 x ULN.
* Adequate hepatic function: total serum bilirubin ≤1.5 x ULN as well as serum AST and ALT ≤1.5 x ULN.
* Subject must be able to participate fully in all aspects of the trial.
* Subject must give voluntary, written consent and HIPAA authorization (US only).

Exclusion Criteria:

* Histologic diagnosis of FAB M3 AML (acute promyelocytic leukemia).
* Clinically active CNS leukemia.
* Known to be HIV positive.
* Prior induction chemotherapy for AML.
* Known active hepatitis B or C or other active liver disease.
* Any major surgery or radiation therapy within 4 weeks prior to study entry.
* Prior cytotoxic chemotherapy within 4 weeks prior to study entry.(Subjects with rapidly rising blast count may be enrolled within 4 weeks of prior cytotoxic chemotherapy).
* Persistent chronic non-hematologic toxicity from prior chemotherapy (other than alopecia) that is > than grade 1.
* Serious concomitant illness (e.g., active pulmonary infection, unstable angina or myocardial infarction within 3 months of study entry, congestive heart failure ≥AHA class 2, stroke within 3 months prior to study entry, uncontrolled hypertension, uncontrolled diabetes, actively bleeding gastric ulcer, etc.).
* Women who are pregnant or lactating.
* History of clinically significant allergic reactions attributed to compounds similar to amonafide or cytarabine.
* Prior enrollment on this trial.
* Any other known condition (familial, sociological, or geographic) or behavior (including substance abuse, psychological or psychiatric illness), which in the investigator's opinion would make the subject a poor candidate for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-08; Study Completion 2009-04

PRIMARY OUTCOMES:
- To determine the rate of complete remission with or without complete hematopoietic recovery (CR + CRi).

SECONDARY OUTCOMES:
Determine the median duration of complete remission with or without complete hematopoietic recovery (CR or CRi)
Determine the proportion of subjects remaining in complete remission (CR +CRi) at 6 months, at 12 months and at 18 months
Determine the median duration of overall survival (OS)
Correlate clinical responses and duration of responses with specific cytogenetic abnormalities
Define the population pharmacokinetic (PK) profile of amonafide and its metabolites when administered as an intravenous infusion daily x 5 days in combination with a standard-dose of cytarabine
Define the safety profile and confirm the acceptability of amonafide and cytarabine
Correlate PK exposure of amonafide and acetylation of amonafide with safety and efficacy assessments in individual subjects

CONTACTS AND LOCATIONS:
Overall Officials: Steven Allen, MD, Principal Investigator — North Shore Hospital
Locations (21):
- United States (19):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - Scripps Cancer Center, San Diego, California
  - University of Colorado Health Sciences Center, Anschutz Cancer Center, Aurora, Colorado
  - University of Florida Health Science Center, Gainesville, Florida
  - Northwestern University, Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - St. Francis Cancer Research Foundation (formerly Indiana Oncology Hematology Consultants and American Health Network of Indiana LLC, Oncology Division), Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - MUSC - Hollings Cancer Center, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - West Virginia University Medical Center, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Regional Cancer Program, London Health Science Center, London, Ontario